CLINICAL TRIAL: NCT02980263
Title: Study of Efficacy and Safety of Canakinumab in Pediatric Patients With Kawasaki Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885D2208
Record Dates: First submitted 2016-10-24; First posted 2016-12-02 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki disease; Coronary artery aneurysm; mucocutaneous lymph node syndrome; lymph node syndrome; canakinumab; intravenous immunoglobulin naïve (IVIG-naïve); intravenous immunoglobulin refractory (IVIG-refractory); pediatric
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Coronary Aneurysm | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kawasaki patients (Experimental)
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab
  Other Names: ACZ885

SUMMARY:
The purpose of this trial is to evaluate whether, in Intravenous Immunoglobulin-naïve or refractory patients diagnosed with active Kawasaki disease, administration of canakinumab controls fever and acute phase reactants.

ELIGIBILITY:
Key Inclusion Criteria:

-Active Kawasaki disease defined as:

* fever ≥38.5°C for ≥5 days
* four out of five of the following criteria: (i) conjunctival injection, (ii) oral mucous membrane changes, (e.g., injected pharynx, or strawberry tongue), (iii) erythema of hands or feet, (iv) polymorphous rash, (v) cervical lymphadenopathy

Key Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study:

* Previous Kawasaki Disease diagnosis, refractory and/or incomplete Kawasaki disease (for IVIG-naïve patients, Cohort 1)
* Patients who had fever for longer than a week (for Intravenous Immunoglobulin-naïve patients, Cohort 1), or longer than 14 days (for Intravenous Immunoglobulin-refractory patients, Cohort 2)
* History of hypersensitivity to any of the study drugs or to drugs or similar chemical classes or excipients (e.g. citric acid and anhydrous sodium chloride disodium edetate dehydrate polysorbate 80; sodium hydroxide; water for injections)

Other protocol-defined inclusion/exclusion may apply.

Ages: 28 Days to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-11-15 (Estimated); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
resolution of fever | Day 3/4

SECONDARY OUTCOMES:
proportion of patients with C-reactive Protein reduction | 12 weeks
proportion of patients developing coronary artery aneurysms | 12 weeks
time to resolution of fever | 12 weeks
proportion of patients with remittent fever | 12 weeks
size of coronary artery aneurysm | 24 weeks
Coronary artery aneurysm evolution over time | 12 weeks
proportion of patients with coronary artery aneurysm | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Undecided